CLINICAL TRIAL: NCT05467787
Title: Comparing Message-based Psychotherapy to Once-weekly, Video-based Psychotherapy for Moderate Depression and Anxiety: A Pilot Study
Brief Title: Comparing Message-based Psychotherapy to Once-weekly, Video-based Psychotherapy for Moderate Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Talkspace (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Thomas Derrick Hull, Research Director, Talkspace
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007239
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Message-based psychotherapy (MBP) (Experimental)
  Interventions: Behavioral: Message-based psychotherapy (MBP)
- Video-chat psychotherapy (VCP) (Experimental)
  Interventions: Behavioral: Video-chat Psychotherapy (VCP)

INTERVENTIONS:
Behavioral: Message-based psychotherapy (MBP) — Message-Based Psychotherapy (MBP) allows patients to chat with an assigned licensed therapist as frequently as they wish. After consumers complete an intake and select a therapist, the consumer can begin chatting with their therapist right away, and as often as they wish. Therapists respond to text within 15 minutes to an hour during office hours, and within 14 hours outside of office hours. Thus, MBP is not fully synchronous. This enables therapists to deliver care to a larger number of patients than is possible under synchronous methods by disentangling the therapist's time from the patient's time to respond. It also has the potential to improve quality as it gives the therapist time to think through the most effective response and intervention. MBP will be based on CBT, PST or IPT intervention strategies.
  Arms: Message-based psychotherapy (MBP)
Behavioral: Video-chat Psychotherapy (VCP) — Video Chat Only (VCP) consists of weekly psychotherapy appointments that last between 30-45 minutes. These sessions are conducted using Agora, a secure, HIPAA-compliant video conferencing service that is seamlessly integrated into the Talkspace platform application. Therapists will provide evidence-based treatments for depression and anxiety.
  Arms: Video-chat psychotherapy (VCP)

SUMMARY:
This study is concerned with evaluating an innovative care delivery platform that is becoming widely available but has not been adequately evaluated in a clinical trial. Primarily, this study is concerned with whether text based care is clinically effective, and if that effect is a function of (1) intervention intensity, (2) timeliness and match of therapeutic recommendations and (3) more stable mood and function over time. Based on the existing, yet limited data in the field, there is evidence to suggest that more frequent encounters with a psychotherapist results in better treatment adherence and faster and more stable response to treatment.

DETAILED DESCRIPTION:
Mobile psychotherapies have been shown to be reliable and effective platforms for delivering evidence-based psychotherapies, and have the potential to reach millions of lives. Several recent randomized clinical trials demonstrate that mobile psychotherapy is effective for mild to moderate depression. These studies also demonstrate that mobile psychotherapy overcomes transportation, time, and stigma barriers for minority and rural individuals. These interventions are found to be culturally relevant and avoid the stigma concerns faced by many minorities and immigrant populations and improve access for those who are too physically disabled to leave home for in-person treatment. Available platforms range from fully self-guided treatment, text-based care, and telephone based psychotherapy. Although self-guided care may be the most cost efficient method of care, recent research shows that this is a highly under-utilized form of care and in soon to be released publication from our group, most patients find this a less appealing form of treatment because of the lack of accountability of the treatment and motivational issues that are a consequence of these illnesses. Indeed, other work suggests that consumer internal resources such as motivation fatigue and illness burden impact engagement with self-guided treatment. Although there is a population to which self-guided treatment may be appealing, in the broader context, access to a coach or expert is needed for these to be effective models of care.

Text-based care however is becoming a widely popular and available form of psychotherapy delivery. Part of the appeal of text-based care is that consumers can access care when they need and at their convenience, and may be able to have more frequent contact with their therapists over the course of treatment. Telephone based psychotherapy is a well-established form of psychotherapy delivery, with several meta-analyses demonstrating not only clinical equivalency with face-to-face psychotherapy, but better adherence to treatment. However, most telephone-based psychotherapy is delivered in a traditional manner, with one-hour, weekly appointments. Although this is an effective manner of care, it still requires that consumers set aside time during the week to receive care and does not allow for in-the-moment care.

Conceptually, text-based care has many potential therapeutic advantages over traditionally delivered telephone-based care. This model of care is similar to Ecological Momentary Intervention (EMI). This intervention model is based on the theory that interventions have their biggest clinical impact when the consumer is at their greatest level of receptivity, and through better timing and tailoring, improve the consumer's readiness to change, self-efficacy to implement the intervention and great behavioral activation in goal directed behavior.

This study is concerned with evaluating an innovative care delivery platform that is becoming widely available but has not been adequately evaluated in a clinical trial. Primarily, this study is concerned with whether text based care is clinically effective, and if that effect is a function of (1) intervention intensity, (2) timeliness and match of therapeutic recommendations and (3) more stable mood and function over time. Based on the existing, yet limited data in the field, there is evidence to suggest that more frequent encounters with a psychotherapist results in better treatment adherence and faster and more stable response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 19 years old or older
* PHQ-9 score of at least 10 and no more than 20
* Must have a valid email address
* Must be willing to receive assessment survey links via email

Exclusion Criteria:

* Non-English speaking
* Under the age of 19
* PHQ-9 score below 10 or above 20
* Inability to receive emails
* Inability or unwilling to receive assessment survey links via email

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-02-08 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) | Change from Baseline PHQ-9 each week for 12 weeks after treatment starts and at 6 months after treatment starts
  The PHQ-9 consists of 9 depression items and one disability item. Each time is associated with a symptom of depression, which the participant rates whether or not they have experienced the symptom over the last two weeks, with severity rating of 0-3. It is one of the few measures that is brief (it takes less than one minute to give) and has been found to have excellent sensitivity to change over time.
Change in Generalized Anxiety Disorder (GAD-7) | Change from Baseline GAD-7 each week for 12 weeks after treatment starts and at 6 months after treatment starts
  To assess for co-occurring anxiety, we will use the GAD-7, a 7- item screener for generalized anxiety. It consists of items related to GAD. Participants rate on a scale of 0-3 how much they have experienced in the last two weeks. The scale is a valid screener for GAD.

CONTACTS AND LOCATIONS:
Overall Officials: Derrick Hull, PhD, Principal Investigator — Talkspace
Locations (1):
- Talkspace, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Quantitative data is available upon reasonable request with a fully executed Data Use Agreement with Talkspace.

REFERENCES:
- [Derived] Song J, Litvin B, Allred R, Chen S, Hull TD, Arean PA. Comparing Message-Based Psychotherapy to Once-Weekly, Video-Based Psychotherapy for Moderate Depression: Randomized Controlled Trial. J Med Internet Res. 2023 Jun 29;25:e46052. doi: 10.2196/46052. PMID 37384392